CLINICAL TRIAL: NCT03181308
Title: A Phase 1b Dose-Escalation Study of Carotuximab (TRC105) in Combination With Nivolumab in Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Carotuximab (TRC105) Plus Nivolumab in Patients With Metastatic NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105LC102
Record Dates: First submitted 2017-06-01; First posted 2017-06-08 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — carotuximab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TRC105 plus Nivolumab (Experimental)
  Interventions: Drug: Carotuximab (TRC105); Drug: OPDIVO

INTERVENTIONS:
Drug: Carotuximab (TRC105) — Anti Endoglin Antibody
  Other Names: TRC105
Drug: OPDIVO — Programmed Death Receptor-1
  Other Names: Nivolumab

SUMMARY:
This is a multi-center, open-label, nonrandomized, dose-escalation, Phase 1b study of carotuximab in combination with standard dose nivolumab in patients with NSCLC that has progressed on or after platinum-based chemotherapy or PD-1/PD-L1 checkpoint inhibition, as a single agent or with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic non-small cell lung cancer (NSCLC) with disease recurrence or progression during or after prior platinum-containing doublet chemotherapy regimen
2. Histologically confirmed metastatic non-small cell lung cancer (NSCLC) that has relapsed following prior PD-1/PD-L1 checkpoint inhibitor therapy without Grade 3 immune-related toxicity, which may or may not have included concurrent chemotherapy. Relapse following prior PD-1 checkpoint therapy is defined as confirmed progressive disease following stable disease or better (e.g., iSD, iPR, iCR) on at least 1 tumor assessment.
3. Patients with an active oncogenic driver (e.g., epidermal growth factor [EGFR], activin-receptor-like kinase 1 [ALK1], or the proto-oncogene tyrosine-protein kinase ROS-1) must have progressed on or after a US Food and Drug Administration (FDA)-approved therapy for that aberration
4. Patients who received adjuvant or neoadjuvant platinum-doublet chemotherapy (after surgery and/or radiation therapy) and developed recurrent or metastatic disease within 6 months of completing therapy are eligible.
5. Patients with recurrent disease > 6 months after adjuvant or neoadjuvant platinum-based chemotherapy, who also subsequently progressed during or after a platinum- doublet regimen given to treat the recurrence, are eligible.
6. Formalin fixed, paraffin-embedded (FFPE) tumor tissue block that permits the preparation of 20 unstained slides of tumor sample (archival) - Biopsy must be excisional, incisional, or core. Needle aspiration is insufficient. In cases where archival tumor tissue is unavailable, tumor biopsy will be required prior to treatment initiation.
7. Programmed death ligand 1 (PD-L1) determination by validated immunohistochemistry assay
8. Measurable disease by iRECIST
9. Age ≥ 18 years
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
11. Resolution of all acute adverse events resulting from prior cancer therapies to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤ 1 or baseline (except alopecia or neuropathy)
12. Adequate organ function
13. Willingness and ability to consent for self to participate in study
14. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Autoimmune disease requiring treatment within the past twelve months.
2. Condition requiring systemic treatment with either corticosteroids
3. History or active interstitial lung disease
4. Prior therapy with T-cell therapy, including an immune checkpoint inhibitor. Patients who received prior immune checkpoint inhibitor therapy are allowed in Expansion Cohort 2 in the absence of recurrent grade 2 (except skin, endocrine and constitutional symptoms), or ≥ 3 immune-related toxicity).
5. Prior treatment with carotuximab
6. Current treatment on another therapeutic clinical trial
7. Receipt of systemic anticancer therapy, including investigational agents, within 28 days prior to study treatment (Note: If anticancer therapy was given within 28 days prior to starting study treatment, patients are not excluded if ≥ 5 times the elimination half-life of the drug has elapsed.)
8. Major surgical procedure or significant traumatic injury within 4 weeks prior to study treatment, and must have fully recovered from any such procedure; and no date of surgery (if applicable) or anticipated need for a major surgical procedure planned within the next 6 months
9. Chest radiotherapy ≤ 28 days, wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvic bones or equivalent), or limited field radiation for palliation ≤ 14 days prior to study treatment - Such patients must have recovered adequately from any side effects of such therapy.
10. Hypertension defined as blood pressure (BP) systolic > 150 or diastolic > 90 mm Hg (Note: Initiation or adjustment of antihypertensive medication prior to study entry is allowed provided that the average of 3 BP readings prior to study treatment is ≤150/90 mm Hg.)
11. Ascites or pericardial effusion that required intervention within 3 months prior to study treatment
12. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease
13. Angina, myocardial infarction (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack TIA), arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) within 6 months prior to study treatment
14. Deep venous thrombosis within 6 months prior to study treatment, unless the patient is anti-coagulated without the use of warfarin for ≥2 weeks prior to study treatment; in this situation, low molecular weight heparin is preferred
15. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g., hereditary hemorrhagic telangiectasia)
16. Thrombolytic use (except to maintain IV catheters) within 10 days prior study treatment
17. Known active viral or nonviral hepatitis or cirrhosis
18. Any active infection requiring systemic treatment
19. History of hemorrhage or hemoptysis (> ½ teaspoon bright red blood) within 3 months prior to study treatment
20. History of peptic ulcer within the past 3 months prior to study treatment, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days prior to study treatment
21. History of gastrointestinal perforation or fistula in the 6 months prior to study treatment, or while previously on antiangiogenic therapy, unless underlying risk has been resolved (e.g., through surgical resection or repair)
22. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
23. Pregnancy or breastfeeding - Female patients must be surgically sterile (i.e., ≥6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of carotuximab. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to study treatment. Male patients must be surgically sterile or must agree to use effective contraception during the study and for at least 180 days following last dose of study drug (carotuximab or nivolumab, whichever occurs later).
24. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, PhD, Study Director — Medical Monitor
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TRACON Pharmaceuticals — http://www.traconpharma.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 8 mg/kg TRC105 + Nivolumab: Dose Level 1 8 mg/kg TRC105 + Nivolumab
  Carotuximab (TRC105): Anti Endoglin Antibody
  OPDIVO (Nivolumab): Programmed Death Receptor-1
- 10 mg/kg TRC105 + Nivolumab: Dose Level 2 10 mg/kg TRC105 + Nivolumab
  Carotuximab (TRC105): Anti Endoglin Antibody
  OPDIVO (Nivolumab): Programmed Death Receptor-1
Period: Overall Study
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
Started | 3 | 8
Completed | 3 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 8 mg/kg TRC105 Plus Nivolumab: Dose Level 1 8 mg/kg TRC105 + Nivolumab Carotuximab (TRC105): Anti Endoglin Antibody OPDIVO (Nivolumab): Programmed Death Receptor-1
- 10 mg/kg TRC105 Plus Nivolumab: Dose Level 2 10 mg/kg TRC105 + Nivolumab Carotuximab (TRC105): Anti Endoglin Antibody OPDIVO (Nivolumab): Programmed Death Receptor-1
- Total: Total of all reporting groups
Arm/Group | 8 mg/kg TRC105 Plus Nivolumab | 10 mg/kg TRC105 Plus Nivolumab | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Continuous [Mean (Full Range); unit: years] | 58 [53 to 67] | 59 [47 to 77] | 59 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 8 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: For DLT evaluation, severity (grade) was classified according to common terminology criteria for adverse events version 4.03 (CTCAE v4.03). DLTs were defined as grade 4 neutropenia persisting for ≥ 5 days, Febrile neutropenia: Grade 4 neutropenia with fever >38.5ºC both sustained over a ≥24-hour period, neutropenic infection (grade ≥ 3 neutropenia with grade ≥ 3 infection), anemia ≥ grade 4, Grade ≥4 thrombocytopenia or Grade ≥3 thrombocytopenia with Grade ≥3 hemorrhage, or grade 3 or 4 nonhematologic toxicity with the following exceptions: asymptomatic electrolyte abnormality that is corrected to Grade 1 or better in <72 hours, grade 3 headache lasting <48 hours. See protocol for Immune related DLT criteria.
Time Frame: Approximately 2-8 months
Population: All patients who received at least a portion of a dose of any study drug (TRC105, Nivolumab)
Measure: Count of Participants; unit: Participants
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
Number analyzed (Participants) | 3 | 8
Participants
  Patients with DLT at 8 mg/kg | 0 | 0
  Patients without DLT at 8 mg/kg | 3 | 0
  Patients with DLT at 10 mg/kg | 0 | 0
  Patients without DLT at 10 mg/kg | 0 | 8

2. Secondary Outcome: Response Rate
Description: Preliminary evidence of antitumor activity of carotuximab (TRC105) plus nivolumab will be evaluated, by assessing response rate and progression-free survival. The best response was measured to iRECIST by MRI or CT scans for each patient with measurable disease who received at least 1 dose of study drug.
Time Frame: Approximately 2-8 months
Population: Number of patients with a baseline scan and at least 1 on study scan were evaluable for response rate determination. Patients were scanned at baseline and every 8 weeks to determine disease status.
Measure: Number; unit: participants
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
Number analyzed (Participants) | 3 | 7
participants
  iSD (Immune Stable Disease) Best Response | 0 | 4
  iPR (Immune Partial Response) Best Response | 1 | 0
  iPD (Immune Progressive Disease) Best Response | 0 | 0
  iCR (Immune Complete Response) Best Response | 0 | 0
  iUPD (Unconfirmed Immune PD) Best Response | 2 | 3

3. Secondary Outcome: Trough Carotuximab (TRC105) Concentrations
Description: Trough (pre-dose) serum carotuximab (TRC105) concentrations will be measured using validated ELISA methods.
Time Frame: 8 weeks
Population: All patients who received at least a portion of a dose of TRC105 with PK samples collected at baseline and at least 1 time point on study. 6 patients had PK analysis completed.
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
Number analyzed (Participants) | 3 | 3
ng/ml | 65233 [46400 to 82700] | 93600 [72600 to 121000]

4. Secondary Outcome: Development of Immunogenicity Antibodies
Description: Number of Participants with carotuximab (TRC105) anti-product antibodies (APA)
Time Frame: Approximately 2-8 months
Population: Anti-product antibody concentrations will be measured using validated ELISA methods. Anti-product antibody concentrations will be evaluated in the context of pharmacokinetic parameters and AE profiles.
Measure: Count of Participants; unit: Participants
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
Number analyzed (Participants) | 3 | 3
Participants
  Ptn with low titer treatment emergent ADA | 0 | 0
  Ptn without treatment emergent ADA | 3 | 3

5. Secondary Outcome: Trough Nivolumab Concentrations
Description: Trough (pre-dose) serum nivolumab concentrations will be measured using validated ELISA methods.
Time Frame: Approximately 2-8 months
Population: All patients who received at least a portion of a dose of TRC105 with PK samples collected at baseline and at least 1 time point on study. Only Cycle 2 Day 1 trough mean serum TRC105 concentrations were analyzed before study closure.
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
Number analyzed (Participants) | 3 | 3
ng/ml | 65233 [46400 to 82700] | 93600 [72600 to 121000]

ADVERSE EVENTS:
Time Frame: From screening until completion of follow-up, on average 6 months
Arm/Group | 8 mg/kg TRC105 + Nivolumab | 10 mg/kg TRC105 + Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/8
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg TRC105 + Nivolumab (N=3) | 10 mg/kg TRC105 + Nivolumab (N=8)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (2)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular access complication (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg TRC105 + Nivolumab (N=3) | 10 mg/kg TRC105 + Nivolumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (6) | 1 (2)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (8) | 1 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 6 (8)
Migraine (Nervous system disorders) | 2 (4) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 3 (3)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03181308/Prot_SAP_000.pdf